CLINICAL TRIAL: NCT04353414
Title: Transmuscular Quadratus Lumborum Block Plus Pericapsular Injection vs Pericapsular Injection for Patients Undergoing Primary Hip Arthroscopy
Brief Title: Transmuscular Quadratus Lumborum Block Plus Pericapsular Injection vs Pericapsular Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20-00058
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Hip Pain Chronic
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular Injection (PCI) group (Active Comparator): Subjects in PCI group will receive the injection through both hip portals administered by the surgeon. 10 mL of 0.25% Bupivacaine Hydrochloride (HCL) will be injected through the anterolateral portal while the additional 10 mL will be injected through the mid-anterior portal.
  Interventions: Procedure: Pericapsular injection; Drug: Bupivacaine Hydrochloride
- Transmuscular QL Block + Pericapsular Injection (PCI) group (Active Comparator): Subjects in the TQLB group will receive the TQLB containing 30mL of 0.5% Bupivacaine Hydrochloride (HCL) plus PCI containing 20 mL of 0.25% of Bupivacaine Hydrochloride (HCL). For PCI, subjects will receive the injection through both hip portals administered by the surgeon. 10 mL of 0.25% Bupivacaine Hydrochloride (HCL) will be injected through the anterolateral portal while the additional 10 mL will be injected through the mid-anterior portal.
  Interventions: Procedure: Transmuscular Quadratus Lumborum Block; Procedure: Pericapsular injection; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Procedure: Transmuscular Quadratus Lumborum Block — Transmuscular Quadratus Lumborum Block (TQLB) is a relatively new block that targets thoracic and lumbar nerves. The decrease in sensation means a decrease in pain. The TQL block will be preformed in addition to an incision-site injection (on hip), called pericapsular injection. The potential risks associated with the Transmuscular Quadratus Lumborum Block (TQLB) include nerve damage and infection at injection site. In addition, there can be temporary sensory and motor loss, depending on the dosage, site of injection and duration of the nerve block. However, the amount (30mL) used in this study meets FDA dosage-regulations for this medication.
  Arms: Transmuscular QL Block + Pericapsular Injection (PCI) group
Procedure: Pericapsular injection — Pericapsular injection (PCI) of 20 mL of 0.25% Bupivacaine HCL (numbing medication) into the incision-site (hip portal sites) to decrease sensation. The potential risks associated with the pericapsular injection include bleeding, infection at injection site and local anesthetic toxicity however, the likelihood is low due to the expertise of the surgeon preforming the injection and the sterile environment and good clinical practice from clinicians, which reduces the likelihood of infection.
Drug: Bupivacaine Hydrochloride — Bupivacaine used for this study is the standard of care for both TQLB and PCI. Pericapsular injection (PCI) contains 10 mL of 0.25% Bupivacaine HCL which will be injected through the anterolateral portal while the additional 10 mL will be injected through the mid-anterior portal.

SUMMARY:
The purpose of this research study is to compare two different treatment options on their effectiveness to reduce post-operative pain, narcotic (opioid pain medication) usage and recovery time in patients undergoing primary hip arthroscopy surgery.

The first treatment option is a Transmuscular Quadratus Lumborum (TQL) block plus hip incision site (Pericapsular) Injection. The TQL block is an ultrasound guided injection between the quadratus lumborum and the psoas muscles in the back. The anesthesiologist will perform the TQL block The second treatment option is only a hip incision site (Pericapsular) Injection. In this group, the surgeon will inject local anesthetic into the incision or hip portal sites to decrease sensation.

DETAILED DESCRIPTION:
This is a phase IV, randomized, single-blind, single-center study comparing postoperative pain, opioid usage and Post-Anesthesia Care Unit (PACU) recovery time for patients who receive a Transmuscular Quadratus Lumborum block (TQLB) plus pericapsular injection versus pericapsular injection (PCI) undergoing primary hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age
* Patients undergoing Primary Hip Arthroscopy
* Patients diagnosed with femoroacetabular impingement (FAI)
* Patients who consent to be randomized.

Exclusion Criteria:

* Patients younger than 18 and older than 65;
* Patients with a history of chronic pain that have used opioids for pain management for 3 months or longer;
* Patients with diagnosed or self-reported cognitive dysfunction;
* Patients with a history of neurologic disorder that can interfere with pain sensation;
* Patients with a history of drug or recorded alcohol abuse;
* Patients who are unable to understand or follow instructions;
* Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
* Patients with an allergy or contraindication to any of the medications used in the study, or patients with a contraindication to any study procedures;
* Patients with BMI over 40;
* Any patient that the investigators feel cannot comply with all study related procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Comparison of post-operative pain as per the Visual Analogue Scale (VAS) | 1 Day of surgery
  This will be measured by using Visual Analogue Scale (VAS) pain scores and compared between the 2 treatment groups after surgery. The distribution of pain Visual Analogue Scale (VAS) scores in post- surgical patients will describe their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain Visual Analogue Scale (VAS) have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Comparison of post-operative pain as per the McGill pain scores | 1 Day of surgery
  This will be determined by the McGill Pain questionnaire (MPQ) scores and compared between the 2 treatment groups during the post-operative period. The MPQ assesses three separate components of the pain experience: the sensory intensity, the emotional impact and the cognitive evaluation of pain. Each descriptor is ranked on a 0 ("none") to 3 ("severe") intensity scale.

SECONDARY OUTCOMES:
Use of Opioids by participants | 1 Day of surgery
  This will be assessed by the pain medications given to the participants depending on their pain level.
Comparison in Post-Anesthesia Care Unit (PACU) Phase 1 recovery time by treatment group | 1 Day of surgery
  This will be an observation of the time it takes the patient in the immediate post op period to transition to Phase II. Factors such as severe pain and post op nausea and vomiting may affect a patient's Phase I recovery time so the study want to compare this parameter between both treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Uchenna Umeh, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to uchenna.umeh@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.